CLINICAL TRIAL: NCT02745470
Title: Effects of a GLP-1 Receptor Agonist on Functional Activation and Connectivity of the Brain Measured by Functional MRI
Brief Title: Effects of a GLP-1 Receptor Agonist on Functional Activation and Connectivity of the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-1507-038-686
Record Dates: First submitted 2016-04-17; First posted 2016-04-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2016-02

CONDITIONS: Diabetes Mellitus
Keywords: lean/obese diabetes mellitus; functional MRI; GLP-1; appetite; activation of brain; connectivity
MeSH Terms: conditions — Diabetes Mellitus | interventions — lixisenatide; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide injection (Experimental): intervention : Lyxumia® pen injection 10 microgram (Lixisenatide) subcutaneous injection 30 minutes before functional MRI
  Interventions: Drug: Lixisenatide
- Normal saline (Placebo Comparator): control : normal saline 0.3 cc subcutaneous injection before functional MRI
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lixisenatide — Colorless, transparent liquid contained in a glass prefilled syringe pen-like injection (GLP-1 receptor agonist)
  Other Names: Lyxumia® pen injection
  Arms: Lixisenatide injection
Other: Placebo — Normal saline injection before performing fMRI
  Other Names: Normal saline injection
  Arms: Normal saline

SUMMARY:
The aims this study is to explore the effect of a GLP-1 receptor agonist on the degree of brain activation and connectivity obtained by functional magnetic resonance imaging in lean and obese type 2 diabetes

DETAILED DESCRIPTION:
Fifteen lean [BMI(body mass index) less than 23 kg/m2] type 2 diabetes subjects and fifteen obese (BMI more than 26 kg/m2) subjects with type 2 diabetes treated by diet and/or metformin, SU(sulfonylurea), DPP4-inhibitors(Dipeptidyl peptidase-4 inhibitor) will be recruited. Every subject will be studied on 2 separate days in random order with 1-2 week intervals. These participants will be injected either normal saline or 10 mcg of lixisenatide in a cross-over fashion. Neuroimaging composed with resting-12-min, visual stimulation task-12-min, T1-5-min, and diffusion tensor image-12-min will be proceeded. Ad lib buffet will be provided to every participant and the intake will be measured. Surveys about appetite and mood will be done before and after neuroimaging test and buffet eating.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 23kg/m2 or BMI ≥ 26kg/m2
* participants with diabetes treated by diet or oral antidiabetic drug, HbA1c less than 8.5%

Exclusion Criteria:

* Those who diagnosed by Type 1 diabetes
* History of insulin therapy
* Aspartate aminotransferase(AST) or Alanine transaminase(ALT) >2.5 times of upper normal reference range
* Estimated Glomerular Filtration Rate(eGFR) <30 mL/min/1.73m2
* Those who can't be performed MRI

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference of BOLD (Blood oxygenation level-dependent) signal in hypothalamus | 10min (40 min after injection)
Whole brain connectivity | 20min (50 min after injection)

SECONDARY OUTCOMES:
appetite change | -30min, 45min(after fMRI), 70min(after buffet)
  Visual analoge scale-questionnaire consisting of 8 questions (Flint, Raben, Blundell, & Astrup, 2000)
mood change | -30min, 45min(after fMRI), 70min(after buffet)
  Visual analoge scale-questionnaire consisting of 16 questions (Boggieo et al., 2008)
intake of food in the buffet | 50min
  It will be provided quantified juice and milk , boiled eggs, bread , bananas and chocolate bars.
  Participants may eat freely for 20 minutes. Then measure the intake of participants.
  Compares whether the difference in food intake pattern .

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Study Chair — Associate Professor Division of Endocrinology and Metabolism Department of Internal Medicine Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided